CLINICAL TRIAL: NCT00147056
Title: A Study to Evaluate the Safety and Feasibility of Transcranial MRI-Guided Focused Ultrasound Surgery in the Treatment of Brain Tumors
Brief Title: MRI-Guided Focused Ultrasound Feasibility Study for Brain Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT002
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor
Keywords: Brain tumor; Brain Lesions; Brain Cancer; ExAblate
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExAblate transcranial system (Experimental): MR Guided Focused Ultrasound
  Interventions: Device: ExAblate transcranial system

INTERVENTIONS:
Device: ExAblate transcranial system — MRI-Guided Focused Ultrasound Feasibility Study for Brain

SUMMARY:
The purpose of this study is to evaluate the safety of MRI-guided focused ultrasound thermal ablation of brain tumors performed through intact human skull using the ExAblate transcranial system. We will collect data to establish the basic safety of this type of treatment as the basis for later studies that will evaluate its clinical efficacy.

DETAILED DESCRIPTION:
In this non-randomized feasibility study, FUS under MRI-guidance and thermometry will be given through intact human skull to brain tumor in up to ten (10) subjects. These subjects will be followed over a 3-month period with contrast MRI and clinical exams.

The objectives are:

1. To evaluate the safety of ExAblate TcMRgFUS treatment delivered through intact human skull to the brain, during the treatment, and during the follow-up period of 3 months.
2. To evaluate the effect of thermal ablation in the target tumor with contrast MR imaging to identify viable tumor, and non-viable thermally ablated tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women.
2. Age between 18 and 70 years, inclusive.
3. Able and willing to give informed consent.
4. Subjects with (newly diagnosed or recurrent) metastatic cancer for whom surgery, radiation, or radiosurgery has not been advised by the treating physician.
5. The targeted tumor tissue is located in the cerebral hemispheres, > 2.5 cm from the inner table of the skull. Non-targeted parts of the tumor may extend outside the treated tumor limits.
6. Tumor(s) are clearly defined on pre-therapy contrast enhanced MRI scans.
7. Size of the targeted portion of the tumor (i.e. prescribed Region Of Treatment) is less than 2.5 cm in diameter or 8 cm3 in volume. The non-targeted tumor tissue may exceed the targeted volume.
8. Karnofsky rating 70-100 (See Appendix A).
9. ASA score 1-2.
10. Able to communicate sensations during the ExAblate MRGFUS procedure.
11. Able to attend all study visits (i.e. life expectancy of at least 3 months).
12. At least 14 days passed since last brain surgery, or intracranial radiation therapy/radiosurgery

Exclusion Criteria:

1. The subject presents with:

   - Symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papaedema).

   - Unstable hemodynamic status including: i. Documented myocardial infarction within six months of enrollment. ii.Symptomatic coronary artery stenosis. iii. Congestive heart disease requiring medication. iv. Anti-arrhythmic drug medication. v. Cardiac pacemaker. vi. Severe hypertension (diastolic BP > 100 on medication).
2. Anti-coagulant therapy, on medications known to increase risk of hemorrhage, (e.g.: non-steroidal anti-inflammatory drugs (NSAIDs), statins
3. TIA or stroke in the last 1 month
4. Insulin-dependent diabetes mellitus
5. Immunosuppression (corticosteroids to prevent brain edema are permitted)
6. Known sensitivity to gadolinium-DTPA
7. Contraindications to MRI such as non-MRI-compatible implanted devices
8. Large subjects not fitting comfortably into the MRI scanner
9. Difficulty laying supine and still for up to 4 hours in the MRI unit or claustrophobia
10. Untreated, uncontrolled Sleep apnea
11. Positive pregnancy test (for pre-menopausal women)
12. Known life-threatening systemic disease
13. More than 3 metastatic tumors
14. History of abnormal bleeding and coagulopathy
15. Use of Avastin in the preceding two weeks or planned use in the forthcoming two weeks and VEGF inhibitors within + 30 days of treatment
16. Patients with a history of uncontrolled seizures or who are not on anti seizure medication (e.g., Phenytoin 100 mg PO t.i.d. or Keppra 500 mg po bid) before the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Serious and Non-Serious Adverse Events after MRI Guided Focused ultrasound treatment for brain tumors | Up to 3 months
  To evaluate the safety of ExAblate TcMRgFUS treatment delivered through intact human skull to the brain, during the treatment and during the follow-up period of 3 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- See also: Sponsor web page — http://www.insightec.com